CLINICAL TRIAL: NCT00194753
Title: Adjuvant Therapy for High-Risk Localized Breast Cancer With Weekly Adriamycin +/- Oral Cytoxan With Continuous G-CSF Support for 12 Weeks Followed by Weekly Taxol for 12 Weeks, Phase II
Brief Title: Adjuvant Therapy for High-Risk Breast Cancer With Wkly Adriamycin & Oral Cytoxan With G-CSF for 12 Wks; Wkly Taxol x 12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Amgen (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18229-A; 00-5889-A 07 (Other: UW Human Subjects Division)
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Breast Neoplasm
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Doxorubicin; Cyclophosphamide; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Weekly doxorubicin (24 mg/m2 IV) with daily oral cyclophosphamide (60 mg/m2 PO) for 12 weeks with G-CSF support days 2 - 7 of each week followed by weekly paclitaxel (80 mg/m2 IV) for 12 weeks.
  Interventions: Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: G-CSF

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2 IV for 12 weeks following completion of doxorubicin and cyclophosphamide
Drug: Doxorubicin — 24 mg/m2 IV weekly x 12
Drug: Cyclophosphamide — 60 mg/m2 PO daily for 12 weeks
Drug: G-CSF — 5 mcg per kg subcutaneously days 2 - 7 during doxorubicin and cyclophosphamide for 12 weeks

SUMMARY:
The primary objectives of the study are to evaluate the feasibility and toxicity of treatment with 12 weeks of Adriamycin with daily oral Cytoxan with G-CSF support followed by 12 weeks of Taxol. Feasibility will be assessed by comparing the delivered dose intensity of each drug to the delivered dose intensity in previous trials. Toxicity will be assessed by comparing the incidence and severity of toxicity with these drugs to previous trials using these drugs in the same combination. We hypothesize metronomic, dose dense treatment as given in this study will be less toxic and more effective than historical regimens using the same drugs in a less metronomic, dose dense manner.

DETAILED DESCRIPTION:
The systemic cancer treatments used in this study (Adriamycin, Cytoxan and Taxol) are all delivered in a dose dense, metronomic manner (weekly or daily). It is our hypothesis that dose dense treatment will result in optimum delivered dose intensity while minimizing toxicity. We will test these hypotheses by comparing the delivered dose intensity of the drugs to the delivered dose intensity of standard regimens. We will also compare time to relapse, survival and toxicity of this treatment to historic, standard regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically confirmed diagnosis of primary breast carcinoma that has been surgically resected. (This regimen is not intended for neoadjuvant treatment.)
* The attending physician must judge the patient to be an appropriate candidate for Adriamycin based adjuvant chemotherapy. Appropriate candidates generally include those with stage II or III breast cancer. The individual attending physician, however, should make the decision.
* Tumor HER-2/neu expression must be determined prior to study enrollment. Assessment may be by fluorescence in situ hybridization (FISH) assay or by immunocytochemistry (ICC). If determination is "intermediate" by immunocytochemistry, FISH must be performed. Protocol therapy is determined by HER-2/neu result.
* Patient must be at least 18.
* The patient must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* Pre-study hematologic values required for entry onto trial are: WBC greater than= 4,000/mm3, ANC greater than= 1,500/mm3 and platelets greater than= 100,000/mm3.

Exclusion Criteria:

* Patients with significant renal dysfunction (creatinine greater than 1.5 x institutional upper limit of normal (IULN)) or hepatic dysfunction (bilirubin greater than IULN; transaminases greater than 2.5 x IULN) are not eligible.
* Except for the following, no prior malignancy is allowed: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient has been disease free for 5 years.
* Patients with clinically apparent cardiac disease, or history of same, are not eligible. Patients who are > 60 years of age or who have a history of hypertension must have a MUGA prior to enrollment. LVEF must be normal.
* Patients who have received prior chemotherapy or radiotherapy are not eligible.
* Patients who are pregnant or breastfeeding are not eligible. Women of child bearing potential must have a serum pregnancy test that is negative and agree to practice adequate contraception.
* Patients with active infection are not eligible.
* Patients who are known to be infected with HIV, hepatitis B or hepatitis C are not eligible. Testing is not required unless there is a high index of clinical suspicion.
* Patients suffering from psychiatric impairment are not eligible.
* Patients with known hypersensitivity to trimethoprim or sulfonamides are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Delivered dose intensity | 24 weeks
Toxicity | 24 weeks

SECONDARY OUTCOMES:
Time to treatment failure | 7 years
Overall survival | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Georgiana K. Ellis, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington/Seattle Cancer Care Alliance, Seattle, Washington, United States